CLINICAL TRIAL: NCT02693119
Title: A Prospective, Randomized, Double-Masked, Vehicle Controlled, Phase 2 Clinical Study to Evaluate the Safety, Tolerability and Efficacy of Elamipretide Topical Ophthalmic Solution in Subjects With Leber's Hereditary Optic Neuropathy (LHON)
Brief Title: A Study Investigating the Safety, Tolerability, and Efficacy of Elamipretide Topical Ophthalmic Solution for Treatment of Leber's Hereditary Optic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPILH-201
Record Dates: First submitted 2016-02-15; First posted 2016-02-26 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Leber's Hereditary Optic Neuropathy
Keywords: LHON; Ocuvia™; elamipretide; MTP-131
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): One drop elamipretide (MTP-131) 1% topical ophthalmic solution BID applied to the left eye (OS) and one drop of vehicle topical ophthalmic solution BID in the fellow eye
  Interventions: Drug: elamipretide (MTP-131) 1% topical ophthalmic solution; Drug: Vehicle topical ophthalmic solution
- Group 2 (Experimental): One drop elamipretide (MTP-131) 1% topical ophthalmic solution BID applied to the right eye (OD) and one drop of vehicle topical ophthalmic solution BID in the fellow eye
  Interventions: Drug: elamipretide (MTP-131) 1% topical ophthalmic solution; Drug: Vehicle topical ophthalmic solution
- Group 3 (Experimental): One drop elamipretide (MTP-131) 1% topical ophthalmic solution BID applied to both eyes (OU).
  Interventions: Drug: elamipretide (MTP-131) 1% topical ophthalmic solution
- OLE (Experimental): One drop elamipretide (MTP-131) 1% topical ophthalmic solution BID applied to both eyes (OU).
  Interventions: Drug: elamipretide (MTP-131) 1% topical ophthalmic solution

INTERVENTIONS:
Drug: elamipretide (MTP-131) 1% topical ophthalmic solution
  Other Names: MTP-131; Bendavia
Drug: Vehicle topical ophthalmic solution
  Arms: Group 1; Group 2

SUMMARY:
This is a Phase 2, prospective, randomized, double-masked, vehicle controlled, single-center study in approximately 12 subjects with LHON to evaluate safety, tolerability and efficacy of elamipretide (MTP-131) topical ophthalmic solution in this patient population. At the conclusion of 52 weeks of treatment, subjects will be offered the opportunity to enter an Open Label Extension for up to 48 additional weeks of treatment.

DETAILED DESCRIPTION:
This was a prospective, randomized, double-masked (DM), vehicle-controlled, single-center study plus open label extension period (OLE) in which approximately 12 subjects with LHON having the genetic mtDNA mutation m.11778G>A were randomized in a masked manner into 1 of 3 groups in a 1:1:1 ratio: one drop of elamipretide 1.0% topical ophthalmic solution twice daily (BID) in the: left eye, right eye, or both eyes.

After completion of the 52-week treatment period or the Week 56 follow-up period, subjects were invited to participate in the OLE period for up to 108 weeks. During the OLE participants received 1% topical opthalmic elamipretide in both eyes (OU) daily. If a subject did not consent to the OLE, he/she completed the study at the Week 56 (±7 days) visit. There were 4 periods in this study: (1) screening period (up to 6 weeks); (2) double-masked treatment period (52 weeks); (3) OLE period (up to 108 weeks), and (4) follow-up period (4 weeks) after completion of End-of-Treatment (EOT) visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 and ≤ 50 years old at the time of loss of vision in the second eye.
* Able to provide informed consent and willing to comply with all study visits and examinations
* Diagnosis of LHON based on clinical and ophthalmic functional/anatomic test findings, and satisfactory documentation of the mitochondrial DNA mutation m.11778G>A
* Loss of vision in both eyes of ≥1 year and ≤10 years at the time of the Screening Visit and current clinically stable visual function (as assessed by the Investigator)
* Able to self-administer eye drops as demonstrated at screening or having a care provider who can do so
* Documentation of having satisfactorily completed at least two previous Humphrey automated visual field tests prior to screening.
* Women of childbearing potential must agree to use birth control as specified in the protocol from the date they sign the informed consent form

Exclusion Criteria:

* Any other ocular pathology requiring treatment with prescription topical ophthalmic drops (e.g., glaucoma, dry eye)
* Cup to disc ratio of > 0.8 in either eye
* Media opacity, suboptimal pupillary dilatation, or refractive error that interferes with adequate retinal imaging
* Known to be immunocompromised or receiving systemic immunosuppression
* Any disease or medical condition that in the opinion of the Investigator would prevent the subject from participating in the study or might confound study results
* Participation in other investigational drug or device clinical trials within 30 days prior to enrollment, or planning to participate in any other investigational drug or device clinical trials within 30 days of study completion
* Women who are pregnant or lactating

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03; Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Sadun, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Doheny Eye Center, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2: One drop elamipretide (MTP-131) 1% topical ophthalmic solution BID applied to a single eye and one drop of vehicle topical ophthalmic solution BID in the fellow eye
Period: Double-Blind Period
Arm/Group | Group 2 | Group 3
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0
Period: Open-Label Period
Arm/Group | Group 2 | Group 3
Started | 8 | 4
Completed | 8 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants for whom age (continuous) was measured.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 2 | Group 3 | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (14.47) | 30.0 (4.83) | 33.6 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 0 | 7
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 1 | 0 | 1
Elamipretide eye [Count of Participants; unit: Participants]
  right eye only | 4 | 0 | 4
  left eye only | 4 | 0 | 4
  both eyes | 0 | 4 | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.70 (3.937) | 29.43 (2.081) | 26.94 (3.796)

OUTCOME MEASURES:

1. Primary Outcome: Double Masked Period: Incidence of Ocular TEAEs
Description: The incidence of ocular treatment emergent adverse events (TEAEs).
Time Frame: Assessed at each visit: Baseline, Day 5 Visit, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 (End of treatment visit) and Week 56 (Follow up visit)
Population: All participants for whom ocular AEs were measured.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Double Masked Group Vehicle Eyes: 4 participants received vehicle in the left eye only, 4 participants received 1% elamipretide in the right eye only
- Double Masked Group Elamipretide Eyes: 4 participants received 1% elamipretide in the left eye only, 4 participants received 1% elamipretide in the right eye only, 4 participants received 1% elamipretide in both eyes
Arm/Group | Double Masked Group Vehicle Eyes | Double Masked Group Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
eyes
  Conjunctival hyperaemia | 3 | 8
  Punctate keratitis: number analyzed (Participants) | 1 | 12
  Punctate keratitis: number analyzed (eyes) | 1 | 16
  Punctate keratitis | 1 | 3
  Dry eye | 0 | 3
  Eye irritation | 1 | 2
  Eyelid irritation: number analyzed (Participants) | 1 | 12
  Eyelid irritation: number analyzed (eyes) | 1 | 16
  Eyelid irritation | 1 | 2
  Eyelid exfoliation: number analyzed (Participants) | 1 | 12
  Eyelid exfoliation: number analyzed (eyes) | 1 | 16
  Eyelid exfoliation | 1 | 1
  Lacrimation increased | 0 | 2
  Choroidal neovascularisation | 0 | 1
  Conjunctival oedema | 0 | 1
  Eyelid oedema | 0 | 1
  Noninfective conjunctivitis | 0 | 1
  Immune system disorders: Hypersensitivity | 1 | 1
  Infections and infestations Conjunctivitis | 1 | 1
  Injury, poisoning and procedural complications: Foreign body in eye | 0 | 1
  Injury, poisoning and procedural complications: Skin abrasion | 0 | 1
  Investigations: Intraocular pressure increased | 1 | 1
  Nervous system disorders: Parosmia | 0 | 2

2. Primary Outcome: Open Label Extension: Incidence of Ocular TEAEs
Description: Open Label Extension: The incidence of ocular treatment emergent adverse events (TEAEs).
Time Frame: Assessed at Week 68, 84, 100, 116, 132, 148, 152, Week 160/ (End of treatment visit)
Population: All participants for whom ocular AEs were measured. For the ocular AE Injury, poisoning and procedural complications: Fall, the subject fell and had a black eye. For ocular AE Immune system disorders Seasonal allergy, individual reported seasonal allergies affecting vision in both eyes. For General disorders and administration site conditions Application site pain, individuals reported burning in eyes, worsening of vision upon application of vehicle or elamipretide eyes.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Double Masked Group Vehicle Eyes | Double Masked Group Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
eyes
  Eye disorders Cataract nuclear | 1 | 1
  Eye disorders Ocular hyperaemia | 1 | 1
  Eye disorders Dry eye | 1 | 1
  Eye disorders Eye irritation | 2 | 1
  Eye disorders Eyelid irritation | 1 | 1
  Eye disorders Visual acuity reduced | 1 | 1
  Eye disorders Visual impairment | 0 | 2
  Eye disorders Punctate keratitis | 1 | 0
  General disorders and administration site conditions Application site pain (eyes burn, vision worse) | 3 | 5
  Immune system disorders Seasonal allergy (worsening vision in eyes) | 1 | 1
  Injury, poisoning and procedural complications: Corneal abrasian | 1 | 0
  Injury, poisoning and procedural complications: Eye contusion | 0 | 1
  Injury, poisoning and procedural complications: Fall (resulting in black eye) | 0 | 1

3. Primary Outcome: Double Masked Period: Severity of Ocular TEAEs
Description: The severity of ocular treatment emergent adverse events (TEAEs).
Time Frame: as for outcome 1
Population: All participants for whom ocular AEs were measured.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Vehicle Eyes: Mild; Vehicle Eyes: Moderate; Vehicle Eyes: Severe: 4 participants received vehicle in the left eye only, 4 participants received 1% elamipretide in the right eye only
- Elamipretide Eyes: Mild; Elamipretide Eyes: Moderate; Elamipretide Eyes: Severe: 4 participants received 1% elamipretide in the left eye only, 4 participants received 1% elamipretide in the right eye only, 4 participants received 1% elamipretide in both eyes
Arm/Group | Vehicle Eyes: Mild | Vehicle Eyes: Moderate | Vehicle Eyes: Severe | Elamipretide Eyes: Mild | Elamipretide Eyes: Moderate | Elamipretide Eyes: Severe
Number analyzed (Participants) | 8 | 8 | 8 | 12 | 12 | 12
Number analyzed (eyes) | 8 | 8 | 8 | 16 | 16 | 16
eyes
  Conjunctival hyperaemia | 2 | 0 | 0 | 1 | 1 | 0
  Punctate keratitis | 1 | 0 | 0 | 3 | 0 | 0
  Dry eye | 0 | 0 | 0 | 3 | 0 | 0
  Eye irritation | 1 | 0 | 0 | 2 | 0 | 0
  Eyelid irritation | 1 | 0 | 0 | 2 | 0 | 0
  Eyelid exfoliation | 1 | 0 | 0 | 1 | 0 | 0
  Lacrimation increased | 0 | 0 | 0 | 2 | 0 | 0
  Choroidal neovascularisation | 2 | 0 | 0 | 0 | 0 | 1
  Conjunctival oedema | 0 | 0 | 0 | 1 | 0 | 0
  Eyelid oedema | 0 | 0 | 0 | 1 | 0 | 0
  Noninfective conjunctivitis | 0 | 0 | 0 | 0 | 1 | 0
  Immune system disorders: Hypersensitivity | 1 | 0 | 0 | 1 | 0 | 0
  Infections and infestations Conjunctivitis | 0 | 1 | 0 | 0 | 1 | 0
  Injury, poisoning and procedural complications: Foreign body in eye | 0 | 0 | 0 | 1 | 0 | 0
  Injury, poisoning and procedural complications: Skin abrasion | 0 | 0 | 0 | 1 | 0 | 0
  Investigations: Intraocular pressure increased | 0 | 1 | 0 | 0 | 1 | 0
  Nervous system disorders: Parosmia | 0 | 0 | 0 | 2 | 0 | 0

4. Primary Outcome: OLE: Severity of Ocular TEAEs
Description: The severity of ocular treatment emergent adverse events (TEAEs).
Time Frame: Assessed at Week 68, 84, 100, 116, 132, 148, 152, Week 160/ (End of treatment visit)
Population: All participants for whom ocular AEs were measured.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Vehicle to Elamipretide Eyes: Mild; Vehicle to Elamipretide Eyes: Moderate; Vehicle to Elamipretide Eyes: Severe: 4 participants received vehicle in the left eye only, 4 participants received 1% elamipretide in the right eye only
- Elamipretide to Elamipretide Eyes: Mild; Elamipretide to Elamipretide Eyes: Moderate; Elamipretide to Elamipretide Eyes: Severe: 4 participants received 1% elamipretide in the left eye only, 4 participants received 1% elamipretide in the right eye only, 4 participants received 1% elamipretide in both eyes
Arm/Group | Vehicle to Elamipretide Eyes: Mild | Vehicle to Elamipretide Eyes: Moderate | Vehicle to Elamipretide Eyes: Severe | Elamipretide to Elamipretide Eyes: Mild | Elamipretide to Elamipretide Eyes: Moderate | Elamipretide to Elamipretide Eyes: Severe
Number analyzed (Participants) | 8 | 8 | 8 | 12 | 12 | 12
Number analyzed (eyes) | 8 | 8 | 8 | 16 | 16 | 16
eyes
  Eye disorders Cataract nuclear | 5 | 0 | 0 | 6 | 0 | 0
  Punctate keratitis | 1 | 0 | 0 | 0 | 0 | 0
  Dry eye | 1 | 0 | 0 | 1 | 0 | 0
  Eye irritation | 2 | 0 | 0 | 1 | 0 | 0
  Eyelid irritation | 1 | 0 | 0 | 1 | 0 | 0
  Ocular hyperaemia | 1 | 0 | 0 | 1 | 0 | 0
  Visual acuity reduced | 1 | 0 | 0 | 1 | 0 | 0
  Visual impairment | 0 | 0 | 0 | 2 | 0 | 0
  General disorders and administration site conditions Application site pain | 3 | 0 | 0 | 5 | 0 | 0
  Immune system disorders Seasonal allergy | 1 | 0 | 0 | 1 | 0 | 0
  Injury, poisoning and procedural complications Corneal abrasian | 1 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications Eye contusion | 0 | 0 | 0 | 1 | 0 | 0
  Injury, poisoning and procedural complications: Fall | 0 | 0 | 0 | 1 | 0 | 0

5. Primary Outcome: Double Masked Period: Best Corrected Visual Acuity (BCVA)
Description: Double Masked Period: Best corrected visual acuity (BCVA) using the using the Early Treatment Diabetic Retinopathy Study (ETDRS) scale by visit. ETDRS charts present a series of five letters of equal difficulty on each row, with standardized spacing between letters and rows; there is a total of 14 lines (70 letters), with letter size increasing further geometrically and equivalently in every line by a factor of 1.2589 (or 0.1 log unit), moving up the chart. Minimum score of zero, maximum score of 100. Change from baseline: a more negative score is worse outcome, a more positive score is better outcome. A lower score means less letters were read correctly (worse outcome) and a higher score means more letters were read correctly (better outcome).
Time Frame: as for outcome 1
Population: All participants for whom BCVA was measured.
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Double Masked Group Vehicle Eyes | Double Masked Group Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
letters
  Day 5 | -3.1 (9.34) | -0.5 (4.50)
  Week 4 | 0.3 (3.33) | 1.0 (3.54)
  Week 8 | 2.0 (3.02) | 0.5 (5.29)
  Week 12 | 2.8 (5.15) | 0.4 (6.47)
  Week 16 | 3.0 (3.38) | 0.6 (4.06)
  Week 20 | 4.0 (10.42) | 1.7 (4.63)
  Week 24 | 4.1 (9.98) | 2.1 (3.79)
  Week 28 | 5.5 (11.99) | 1.4 (4.99)
  Week 32 | 4.8 (15.54) | 2.7 (7.67)
  Week 36 | 6.6 (11.73) | 1.9 (4.53)
  Week 40 | 2.6 (11.56) | 3.2 (4.40)
  Week 44 | 6.1 (11.85) | 3.5 (5.97)
  Week 48 | 5.1 (16.58) | 4.8 (4.89)
  Week 52 | 4.6 (16.27) | 2.9 (5.45)
  Week 56 (follow up Visit): number analyzed (Participants) | 3 | 3
  Week 56 (follow up Visit): number analyzed (eyes) | 3 | 3
  Week 56 (follow up Visit) | 1.7 (2.89) | 5.3 (4.16)

6. Primary Outcome: Open Label Extension Period: Best Corrected Visual Acuity (BCVA) Using the Using the Early Treatment Diabetic Retinopathy Study (ETDRS) Scale
Description: Open Label Extension Period: Best corrected visual acuity (BCVA) using the using the Early Treatment Diabetic Retinopathy Study (ETDRS) scale by visit. ETDRS charts present a series of five letters of equal difficulty on each row, with standardized spacing between letters and rows; there is a total of 14 lines (70 letters), with letter size increasing further geometrically and equivalently in every line by a factor of 1.2589 (or 0.1 log unit), moving up the chart. Minimum score of zero, maximum score of 100. Change from baseline: a more negative score is worse outcome, a more positive score is better outcome. A lower score means less letters were read correctly (worse outcome) and a higher score means more letters were read correctly (better outcome).
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160 (follow-up visit).
Population: All participants for whom BCVA was measured.
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Groups:
- Vehicle to Elamipretide: 4 participants who received vehicle in left eye during DM period, now received elamipretide. 4 participants who received vehicle in right eye during former DM period, now received elamipretide.
- Elamipretide to Elamipretide: 8 participants who received 1% elamipretide in left or right eye only during DM period, continued to receive 1% elamipretide in the eye. 4 participants who received 1% elamipretide in both eyes during former DM period, continued to receive 1% elamipretide in both eyes.
Arm/Group | Vehicle to Elamipretide | Elamipretide to Elamipretide
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
letters
  Week 68 | 8.5 (14.16) | 6.00 (7.18)
  Week 84 | 10.6 (18.66) | 5.4 (7.70)
  Week 100: number analyzed (Participants) | 8 | 11
  Week 100: number analyzed (eyes) | 8 | 14
  Week 100 | 6.1 (13.86) | 6.1 (6.12)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | -3.5 (6.36) | 2.5 (0.71)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | 11.3 (14.00) | 5.9 (6.71)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | 11.6 (17.04) | 4.3 (8.36)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | 2.8 (2.50) | 2.9 (4.05)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | 1.7 (2.08) | 7.7 (4.16)

7. Secondary Outcome: Double Masked Period: Photopic Negative Response Electroretinography (PhNR-ERG) A-wave Amplitude
Description: Change from baseline in photopic negative response electroretinography (PhNR-ERG) a-wave amplitude by Visit. Photopic negative response electroretinography (PhNR-ERG) assesses retinal cell function. A decrease in the amplitude of the a-wave is associated with worse outcomes. Change from baseline in a-wave amplitude: a more positive number equals a decrease in amplitude, and therefore a worse outcome, a more negative number mean a better outcome.
Time Frame: Assessed at each visit from Baseline to Week 56 (follow-up visit), except for Day 5 visit.
Population: All participants for whom photopic negative response electroretinography PhNR-ERG was measured.
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Groups:
- Vehicle Eyes: 4 participants received vehicle in the left eye only, 4 participants received 1% elamipretide in the right eye only
- Elamipretide Eyes: 4 participants received 1% elamipretide in the left eye only, 4 participants received 1% elamipretide in the right eye only, 4 participants received 1% elamipretide in both eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µV
  Week 4 | 0.0 (6.61) | 1.3 (6.81)
  Week 8: number analyzed (Participants) | 7 | 11
  Week 8: number analyzed (eyes) | 7 | 14
  Week 8 | -0.2 (6.92) | 0.5 (7.50)
  Week 12 | -3.5 (11.09) | -3.2 (10.18)
  Week 16 | 1.1 (6.71) | 0.7 (6.30)
  Week 20: number analyzed (eyes) | 8 | 15
  Week 20 | 1.5 (4.64) | 1.1 (4.71)
  Week 24 | 2.0 (6.18) | 2.0 (6.56)
  Week 28 | 0.4 (5.11) | 2.5 (5.80)
  Week 32 | 2.0 (8.18) | 0.3 (5.64)
  Week 36: number analyzed (Participants) | 8 | 11
  Week 36: number analyzed (eyes) | 8 | 14
  Week 36 | -2.5 (11.62) | 0.2 (7.00)
  Week 40 | 2.2 (10.07) | 1.5 (6.28)
  Week 44 | 1.0 (11.05) | 3.2 (6.55)
  Week 48 | 3.4 (8.31) | 2.9 (6.19)
  Week 52 | 2.3 (5.58) | 2.0 (5.16)
  Week 56 (Follow up Visit): number analyzed (Participants) | 3 | 3
  Week 56 (Follow up Visit): number analyzed (eyes) | 3 | 3
  Week 56 (Follow up Visit) | 7.0 (2.93) | 5.1 (8.71)

8. Secondary Outcome: Open Label Extension Period: Photopic Negative Response Electroretinography (PhNR-ERG) A-wave Amplitude
Description: as for outcome 7
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160
Population: All participants for whom photopic negative response electroretinography (PhNR-ERG) was measured.
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Groups:
- Vehicle to Elamipretide Eyes: Double Masked Period 4 participants received vehicle in the left eye only, 4 participants received 1% elamipretide in the right eye only
  Open Label Period: All 12 participants received 1 drop of elamipretide 1.0% topical ophthalmic solution BID instilled into both eyes (Oculus Uterque [OU]).
- Elamipretide to Elamipretide Eyes: Double Masked Period: 4 participants received 1% elamipretide in the left eye only, 4 participants received 1% elamipretide in the right eye only, 4 participants received 1% elamipretide in both eyes
  Open Label Period: All 12 participants received 1 drop of elamipretide 1.0% topical ophthalmic solution BID instilled into both eyes (Oculus Uterque [OU]).
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µV
  Week 68 | 3.2 (9.24) | 4.0 (6.00)
  Week 84: number analyzed (Participants) | 7 | 11
  Week 84: number analyzed (eyes) | 7 | 15
  Week 84 | -7.1 (19.27) | 1.8 (6.81)
  Week 100: number analyzed (Participants) | 6 | 9
  Week 100: number analyzed (eyes) | 6 | 12
  Week 100 | 8.0 (5.69) | 4.9 (4.41)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | 5.3 (3.27) | 3.0 (1.71)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | -2.7 (9.39) | 0.3 (5.93)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | 5.7 (7.07) | 1.4 (3.99)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | 5.4 (8.92) | 1.5 (3.84)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | 2.9 (2.82) | 2.82 (7.60)

9. Secondary Outcome: Double Masked Period: Photopic Negative Response Electroretinography (PhNR-ERG) B-wave Amplitude
Description: Change from baseline in photopic negative response electroretinography (PhNR-ERG) b-wave amplitude by visit. Photopic negative response electroretinography (PhNR -ERG) assesses retinal cell function. A decrease in the amplitude of the b-wave is associated with worse outcomes. Change from baseline in b-wave amplitude: a more negative number equals a decrease in amplitude, and therefore a worse outcome, a more positive number mean a better outcome.
Time Frame: Assessed at each visit from Baseline to Week 56 (follow-up visit), except for Day 5 visit.
Population: All participants for whom PhNR-ERG was measured.
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µV
  Week 4 | -9.1 (14.36) | -4.5 (31.48)
  Week 8: number analyzed (Participants) | 7 | 11
  Week 8: number analyzed (eyes) | 7 | 14
  Week 8 | -4.6 (21.82) | -3.4 (22.33)
  Week 12 | 3.5 (17.85) | 14.6 (27.23)
  Week 16 | -2.8 (28.02) | -2.6 (19.83)
  Week 20: number analyzed (eyes) | 8 | 15
  Week 20 | -2.2 (22.48) | -6.4 (29.35)
  Week 24 | -8.9 (20.58) | -1.0 (28.06)
  Week 28 | -0.7 (19.04) | -11.6 (17.75)
  Week 32 | -5.6 (13.57) | 1.8 (24.58)
  Week 36: number analyzed (Participants) | 8 | 11
  Week 36: number analyzed (eyes) | 8 | 14
  Week 36 | 2.4 (29.87) | 2.2 (22.06)
  Week 40 | -0.1 (23.58) | -8.1 (23.17)
  Week 44 | 1.9 (21.35) | -5.0 (21.01)
  Week 48 | -6.9 (24.08) | -10.5 (23.80)
  Week 52 | -1.3 (13.97) | -5.4 (18.99)
  Week 56 (Follow up): number analyzed (Participants) | 3 | 3
  Week 56 (Follow up): number analyzed (eyes) | 3 | 3
  Week 56 (Follow up) | -18.4 (28.05) | -17.5 (49.57)

10. Secondary Outcome: Open Label Extension Period: PhNR-ERG B-wave Amplitude
Description: Change from baseline in photopic negative response electroretinography (PhNR-ERG) b-wave Amplitude by Visit. Photopic negative response electroretinography (PhNR -ERG) assesses retinal cell function. A decrease in the amplitude of the b-wave is associated with worse outcomes. Change from baseline in b-wave amplitude: a more negative number equals a decrease in amplitude, and therefore a worse outcome, a more positive number means a better outcome.
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160
Population: All participants for whom PhNR-ERG was measured.
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µV
  Week 68 | -15.4 (25.98) | -7.4 (17.10)
  Week 84: number analyzed (Participants) | 7 | 11
  Week 84: number analyzed (eyes) | 7 | 15
  Week 84 | -6.0 (23.97) | -13.1 (20.97)
  Week 100: number analyzed (Participants) | 6 | 9
  Week 100: number analyzed (eyes) | 6 | 12
  Week 100 | -28.7 (23.23) | -19.9 (18.04)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | -17.7 (5.23) | -14.2 (4.62)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | 17.1 (44.40) | 4.9 (18.79)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | -17.1 (17.08) | -1.3 (18.81)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | -13.1 (30.88) | -7.3 (18.84)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | -17.8 (14.15) | -38.1 (25.20)

11. Secondary Outcome: Double Masked Period: PhNR Amplitude
Description: Double Masked Period: Change from baseline in PhNR Amplitude by Visit. Photopic negative response electroretinography (PhNR -ERG) assesses retinal cell function. A decrease in PhNR amplitude means worse outcome. Change from baseline: A more negative number means a better outcome, a more positive number means a worse outcome.
Time Frame: Assessed at each visit from Baseline to Week 56 (follow-up visit), except for Day 5 visit.
Population: All participants for whom PhNR Amplitude was measured.
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µV
  Week 4 | -6.4 (22.27) | 0.3 (22.05)
  Week 8: number analyzed (Participants) | 7 | 11
  Week 8: number analyzed (eyes) | 7 | 14
  Week 8 | -4.6 (26.80) | -3.3 (27.28)
  Week 12 | -11.6 (26.59) | -0.7 (14.90)
  Week 16 | -4.5 (10.26) | -3.1 (17.35)
  Week 20: number analyzed (eyes) | 8 | 15
  Week 20 | 0.5 (20.65) | -3.1 (19.58)
  Week 24 | -4.3 (21.51) | -0.5 (16.15)
  Week 28 | -7.1 (26.32) | -1.5 (13.92)
  Week 32 | -4.1 (25.11) | -3.1 (13.61)
  Week 36: number analyzed (Participants) | 8 | 11
  Week 36: number analyzed (eyes) | 8 | 14
  Week 36 | -8.5 (24.94) | -3.4 (10.17)
  Week 40 | -2.3 (23.16) | -4.4 (10.92)
  Week 44 | -9.8 (29.75) | -1.5 (11.91)
  Week 48 | -2.8 (22.76) | -3.7 (13.14)
  Week 52 | -4.0 (25.41) | -3.3 (11.73)
  Week 56 (Follow up): number analyzed (Participants) | 3 | 3
  Week 56 (Follow up): number analyzed (eyes) | 3 | 3
  Week 56 (Follow up) | -1.6 (16.71) | -5.7 (6.45)

12. Secondary Outcome: Open Label Extension Period: PhNR Amplitude
Description: Open Label Extension Period: Change from baseline in PhNR Amplitude by Visit. Photopic negative response electroretinography (PhNR -ERG) assesses retinal cell function. A decrease in PhNR amplitude means worse outcome. Change from baseline: A more negative number means a better outcome, a more positive number means a worse outcome.
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160
Population: All participants for whom PhNR Amplitude was measured.
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µV
  Week 68 | -7.1 (22.91) | 0.5 (16.60)
  Week 84: number analyzed (Participants) | 7 | 11
  Week 84: number analyzed (eyes) | 7 | 15
  Week 84 | -2.5 (25.45) | -2.2 (11.96)
  Week 100: number analyzed (Participants) | 6 | 9
  Week 100: number analyzed (eyes) | 6 | 12
  Week 100 | 3.3 (16.25) | 1.8 (6.50)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | 3.3 (1.03) | -1.2 (6.72)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | -5.1 (20.89) | 0.4 (9.00)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | -3.6 (20.98) | 0.5 (10.75)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | -4.1 (8.75) | -1.4 (4.23)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | -9.9 (4.31) | -10.0 (11.64)

13. Secondary Outcome: Double Masked Period: PhNR/B-wave Amplitude Ratio
Description: Double Masked Period: Change from baseline in PhNR/b-wave amplitude ratio by Visit. Photopic negative response electroretinography (PhNR assesses retinal cell function. A decrease in PhNR amplitude means worse outcome.
Time Frame: Assessed at each visit from Baseline to Week 56 (follow-up visit), except for Day 5 visit.
Population: All participants for whom PhNR was measured.
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
ratio
  Week 4 | -0.102 (0.2225) | -0.033 (0.2793)
  Week 8: number analyzed (Participants) | 7 | 11
  Week 8: number analyzed (eyes) | 7 | 14
  Week 8 | -0.036 (0.3101) | -0.033 (0.3385)
  Week 12 | -0.113 (0.2415) | 0.019 (0.1721)
  Week 16 | -0.059 (0.1179) | -0.070 (0.2285)
  Week 20: number analyzed (Participants) | 8 | 11
  Week 20: number analyzed (eyes) | 8 | 15
  Week 20 | -0.018 (0.2005) | -0.066 (0.2365)
  Week 24 | -0.052 (0.2080) | 0.014 (0.2131)
  Week 28 | -0.044 (0.2281) | -0.024 (0.1634)
  Week 32 | -0.033 (0.2414) | -0.031 (0.1513)
  Week 36 | -0.104 (0.2479) | -0.013 (0.1795)
  Week 40: number analyzed (Participants) | 8 | 11
  Week 40: number analyzed (eyes) | 8 | 14
  Week 40 | -0.007 (0.2190) | -0.046 (0.1202)
  Week 44 | -0.138 (0.3194) | 0.013 (0.2206)
  Week 48 | -0.020 (0.2366) | -0.059 (0.1533)
  Week 52 | -0.044 (0.2428) | -0.029 (0.1299)
  Week 56 (Follow up): number analyzed (Participants) | 3 | 3
  Week 56 (Follow up): number analyzed (eyes) | 3 | 3
  Week 56 (Follow up) | 0.009 (0.2670) | -0.063 (0.1149)

14. Secondary Outcome: Open Label Extension Period: Change From Baseline by Visit PhNR/b Wave Amplitude Ratio
Description: Open Label Extension Period: Change from baseline by visit PhNR/b Wave Amplitude Ratio by visit. A reduced amplitude ratio equals worse outcome.
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160
Population: All participants for whom PhNR-ERG was measured.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
Ratio
  Week 68 | -0.097 (0.2453) | -0.002 (0.1722)
  Week 84: number analyzed (Participants) | 7 | 11
  Week 84: number analyzed (eyes) | 7 | 15
  Week 84 | -0.021 (0.2678) | -0.041 (0.1207)
  Week 100: number analyzed (Participants) | 6 | 9
  Week 100: number analyzed (eyes) | 6 | 12
  Week 100 | 0.012 (0.1523) | -0.003 (0.0796)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | 0.019 (0.0066) | -0.048 (0.0667)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | -0.034 (0.2112) | 0.000 (0.0971)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | -0.055 (0.1957) | 0.032 (0.2010)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | -0.035 (0.0717) | -0.046 (0.0982)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | -0.155 (0.1075) | -0.212 (0.2211)

15. Secondary Outcome: Double Masked Period: Change From Baseline by Visit PhNR Peak to Trough Adjusted for A-wave Amplitude
Description: Double Masked Period: Change from baseline by visit in PhNR Peak to Trough Adjusted for a-wave Amplitude by Visit. Calculated as (b-wave amplitude - PhNR amplitude)/a-wave amplitude. A reduced amplitude ratio equals worse outcome.
Time Frame: Assessed at each visit from Baseline to Week 56 (follow-up visit), except for Day 5 visit.
Population: All participants for whom PhNR-ERG was measured.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
Ratio
  Week 4 | 0.18 (0.392) | -0.21 (1.100)
  Week 8: number analyzed (Participants) | 7 | 11
  Week 8: number analyzed (eyes) | 7 | 14
  Week 8 | -0.03 (0.655) | 1.08 (4.628)
  Week 12 | 0.08 (0.827) | 0.00 (0.962)
  Week 16 | -0.53 (1.260) | -0.01 (0.862)
  Week 20: number analyzed (eyes) | 8 | 15
  Week 20 | -0.32 (0.992) | 0.10 (1.022)
  Week 24 | -0.35 (0.856) | -0.29 (0.746)
  Week 28 | -0.35 (0.819) | -0.21 (1.358)
  Week 32 | -0.24 (0.820) | -0.15 (0.606)
  Week 36: number analyzed (Participants) | 8 | 11
  Week 36: number analyzed (eyes) | 8 | 14
  Week 36 | -0.05 (0.687) | -0.70 (1.162)
  Week 40 | 0.63 (0.546) | 0.02 (1.123)
  Week 44 | -0.68 (0.438) | -0.66 (1.016)
  Week 48 | -0.61 (0.811) | -0.31 (0.769)
  Week 52 | -0.61 (0.291) | -0.37 (0.403)
  Week 56 (Follow up): number analyzed (Participants) | 3 | 3
  Week 56 (Follow up): number analyzed (eyes) | 3 | 3
  Week 56 (Follow up) | -1.22 (0.114) | -0.87 (0.274)

16. Secondary Outcome: Open Label Extension Period: Change From Baseline by Visit PhNR Peak to Trough Adjusted for A-wave Amplitude
Description: Open Label Extension Period: Change from baseline by visit in PhNR Peak to Trough Adjusted for a-wave Amplitude by Visit. [Calculated by b-wave amplitude - PhNR amplitude)/a-wave amplitude.] Photopic negative response electroretinography (PhNR-ERG) assesses retinal cell function. A decrease in the amplitude of the a-wave is associated with worse outcomes. A reduced amplitude ratio equals worse outcome.
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160
Population: All participants for whom PhNR-ERG was measured.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
Ratio
  Week 68 | -0.31 (1.006) | -0.70 (0.859)
  Week 84: number analyzed (Participants) | 7 | 11
  Week 84: number analyzed (eyes) | 7 | 15
  Week 84 | 0.25 (1.700) | -0.09 (1.050)
  Week 100: number analyzed (Participants) | 6 | 9
  Week 100: number analyzed (eyes) | 6 | 12
  Week 100 | -0.30 (0.591) | -0.13 (0.407)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | -0.10 (0.454) | -0.09 (0.103)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | -0.64 (1.189) | -0.46 (0.673)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | -0.77 (0.831) | -0.38 (0.329)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | -0.91 (0.609) | -0.16 (0.437)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | -0.46 (0.457) | -0.92 (1.027)

17. Secondary Outcome: Double Masked Period: PhNR Peak to Trough Amplitude (Unadjusted) From Baseline
Description: Double Masked Period: Change from baseline in PhNR Peak to Trough Amplitude (Unadjusted) by Visit. Calculated as b-wave amplitude - PhNR amplitude. Photopic negative response electroretinography (PhNR-ERG) assesses retinal cell function. A decrease in amplitude is associated with worse outcomes.
Time Frame: Assessed at each visit from Baseline to Week 56 (follow-up visit), except for Day 5 visit.
Population: All participants for whom PhNR-ERG was measured.
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µV
  Week 4 | -2.72 (24.750) | -4.80 (31.025)
  Week 8: number analyzed (Participants) | 7 | 11
  Week 8: number analyzed (eyes) | 7 | 14
  Week 8 | 0.08 (18.496) | -0.08 (31.421)
  Week 12 | 15.16 (38.016) | 15.38 (33.898)
  Week 16 | 1.70 (32.016) | 0.52 (25.629)
  Week 20: number analyzed (eyes) | 8 | 15
  Week 20 | -2.62 (20.398) | -3.29 (21.498)
  Week 24 | -4.57 (25.171) | -0.54 (30.470)
  Week 28 | 6.38 (26.095) | -10.18 (19.504)
  Week 32 | -1.42 (28.294) | 4.86 (26.750)
  Week 36: number analyzed (Participants) | 8 | 11
  Week 36: number analyzed (eyes) | 8 | 14
  Week 36 | 10.94 (48.051) | 5.57 (26.427)
  Week 40 | 2.22 (43.149) | -3.74 (27.206)
  Week 44 | 11.74 (46.933) | -3.46 (26.042)
  Week 48 | -4.12 (34.581) | -6.86 (28.849)
  Week 52 | 2.73 (19.124) | -2.15 (22.109)
  Week 56 (Follow up): number analyzed (Participants) | 3 | 3
  Week 56 (Follow up): number analyzed (eyes) | 3 | 3
  Week 56 (Follow up) | -16.78 (19.472) | -11.80 (49.865)

18. Secondary Outcome: Open Label Extension Period: PhNR Peak to Trough Amplitude (Unadjusted)
Description: Open Label Extension Period: Change from baseline in PhNR Peak to Trough Amplitude (Unadjusted) by Visit. b-wave amplitude - PhNR amplitude. Photopic negative response electroretinography (PhNR-ERG) assesses retinal cell function. A decrease in the amplitude of the a-wave is associated with worse outcomes.
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160
Population: All participants for whom PhNR-ERG was measured.
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µV
  Week 68 | -8.36 (36.178) | -7.92 (21.402)
  Week 84: number analyzed (Participants) | 7 | 11
  Week 84: number analyzed (eyes) | 7 | 15
  Week 84 | -3.50 (13.206) | -10.90 (22.928)
  Week 100: number analyzed (Participants) | 6 | 9
  Week 100: number analyzed (eyes) | 6 | 12
  Week 100 | -32.02 (23.994) | -21.64 (21.432)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | -21.01 (4.193) | -13.01 (11.340)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | 22.26 (42.352) | 4.52 (22.231)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | -13.56 (27.012) | -1.85 (15.341)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | -8.99 (35.662) | -5.84 (19.242)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | -7.87 (11.415) | -28.17 (31.249)

19. Secondary Outcome: Double Masked: VFQ-39 Composite
Description: Double Masked: Change from baseline in Visual Function Questionnaire (VFQ-39) Composite score by visit. National Eye Institute VFQ-39 measures health-related quality of life in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, peripheral vision, and composite score. For each domain: the lowest and highest possible scores are 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom VFQ-39 was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Single Eye: Participants who received 1% elamipretide in one eye and control (placebo) in paired eye.
- Bilateral Eye: Participants who received 1% elamipretide in both eyes.
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
score on a scale
  Week 52 | 6.1 (5.63) | 5.7 (8.07)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit) | 7.8 (7.02) |

20. Secondary Outcome: Open Label Extension Period: VFQ-39 Composite Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Composite score.National Eye Institute VFQ-39 measures health-related quality of life in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, peripheral vision, and composite score. For each domain: the lowest and highest possible scores are 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom change in VFQ-39 composite score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Groups:
- Single Eye in DM Period: Participants who received 1% elamipretide BID in one eye and control (placebo) BID in paired eye in the DM Period, and then received 1% elamipretide BID in both eyes in the OLE Period.
- Bilateral Eye in DM Period: Elamipretide to Elamipretide Eyes
  DM Period: 4 participants received 1% elamipretide in both eyes in DM Period and continued receiving 1% elamipretide in both eyes in the OLE Period
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 6
score on a scale | 5.6 (11.30) | 13.9 (8.66)

21. Secondary Outcome: Open Label Extension Period: VFQ-39 General Health Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) General Health score. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change from baseline in Visual Function Questionnaire (VFQ-39) General Health score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 6
score on a scale | -6.8 (10.58) | 6.7 (11.55)

22. Secondary Outcome: Double Masked: VFQ-39 General Vision Score
Description: Change from baseline in VFQ-39 General Vision Score. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculate
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom change from VFQ-39 General Health score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 8.1 (8.84) | 1.3 (11.09)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | 3.3 (7.64) |

23. Secondary Outcome: Open Label Extension Period: VFQ-39 General Vision Score
Description: as for outcome 22
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change in Visual Function Questionnaire (VFQ-39) General Vision was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 6
score on a scale | 9.3 (13.36) | 6.7 (11.55)

24. Secondary Outcome: Double Masked: VFQ-39 Ocular Pain Score
Description: Change from baseline in VFQ-39 Ocular Pain score. National Eye Institute VFQ-39 measures health-related quality of life in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, peripheral vision, and composite score. For each domain: the lowest and highest possible scores are 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom change from VFQ-39 General Health score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 1.6 (12.39) | 3.1 (6.25)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | 12.5 (12.50) |

25. Secondary Outcome: Open Label Extension Period: VFQ-39 Ocular Pain Score
Description: Change from baseline in VFQ-39 Ocular Pain score by visit. National Eye Institute VFQ-39 measures health-related quality of life in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, peripheral vision, and composite score. For each domain: the lowest and highest possible scores are 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change in Visual Function Questionnaire (VFQ-39) Ocular Pain was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 6
score on a scale | -16.1 (20.04) | -4.2 (7.22)

26. Secondary Outcome: Double Masked: VFQ-39 Near Activities Score
Description: Change from Baseline in VFQ-39 Near Activities Score from Baseline. National Eye Institute VFQ-39 measures health-related quality of life in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, peripheral vision, and composite score. For each domain: the lowest and highest possible scores are 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom change from VFQ-39 Near Activities score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 3.6 (7.53) | 9.2 (9.41)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | 11.1 (9.62) |

27. Secondary Outcome: Open Label Extension Period: VFQ-39 Near Activities
Description: Change from Baseline in Visual Function Questionnaire (VFQ-39) Near Activities score.. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; score ranges from 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom change in VFQ-39 Near Activities score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 6
score on a scale | 8.5 (11.03) | 16.7 (16.67)

28. Secondary Outcome: Double Masked Period: Mean Retinal Nerve Fiber (RNFL) Layer Thickness
Description: Change from baseline in retinal nerve fiber layer thickness by spectral domain optical coherence tomography (SD-OCT). RNFL measures the loss of retinal ganglion cell axons. RNFL thickness decreases as disease progresses. A positive number, or, absence of change from baseline reflects a good clinical outcome, a negative number reflects loss of thickness, or a bad outcome.
Time Frame: Assessed at Baseline and Week 52 (end-of-treatment visit)
Population: All participants for whom Retinal Nerve Fiber Layer Thickness was measured.
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µm | -3.8 (7.52) | -2.6 (4.76)

29. Secondary Outcome: Open Label Extension Period: Retinal Nerve Fiber Layer Thickness
Description: Open Label Extension Period: Change from baseline in Retinal Nerve Fiber Layer Thickness by SD-OCT by visit. Change from baseline in retinal nerve fiber layer thickness by spectral domain optical coherence tomography (SD-OCT). RNFL measures the loss of retinal ganglion cell axons. RNFL thickness decreases as disease progresses. A positive number, or, absence of change from baseline reflects a good clinical outcome, a negative number reflects loss of thickness, or a bad outcome.
Time Frame: Assessed at Baseline, Week 148
Population: All participants for whom Change in Retinal Nerve Fiber Layer Thickness by SD-OCT was measured.
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: eyes
Groups:
- Vehicle to Elamipretide Eyes: Double Masked Period 4 participants received vehicle in the left eye only, 4 participants received vehicle in the right eye only.
  Open Label Period: All 8 participants received 1 drop of elamipretide 1.0% topical ophthalmic solution BID instilled into both eyes (Oculus Uterque [OU]).
- Elamipretide to Elamipretide Eyes: DM Period: 4 participants received 1% elamipretide BID in the left eye only, 4 participants received 1% elamipretide BID in the right eye only, 4 participants received 1% elamipretide BID in both eyes.
  OLE Period: All 8 participants received 1 drop of elamipretide 1.0% topical ophthalmic solution BID instilled into both eyes (Oculus Uterque [OU]).
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 1 | 5
Number analyzed (eyes) | 1 | 3
µm | -1.0 | 1.4 (2.70)

30. Secondary Outcome: Double Masked Period: Visual Field Mean Deviation as Measured by Humphrey Automated Visual Field Testing Stimulus III
Description: Change from Baseline in visual field Mean Deviation(MD) as measured by Humphrey automated visual field testing stimulus III by visit. The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. Mean deviation (MD) is the mean deviation in the patient's results compared to those expected from the age-matched normative database. Lower/More negative scores mean worse outcome, higher/more positive score means better outcome.
Time Frame: Assessed at each visit from Baseline to Week 56 (follow-up visit), except for Day 5 visit.
Population: All participants for whom Visual Field Mean Deviation as Measured by Humphrey Automated Visual Field Testing Stimulus III was measured
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
dB
  Week 4 | 1.1 (3.62) | 2.1 (3.94)
  Week 8 | 0.5 (3.88) | 1.6 (3.82)
  Week 12 | 0.4 (3.85) | 0.9 (3.42)
  Week 16 | 0.3 (1.87) | 1.9 (2.62)
  Week 20 | -0.4 (5.31) | 2.1 (4.23)
  Week 24 | 2.0 (3.33) | 1.1 (2.74)
  Week 28 | 1.7 (4.40) | 1.3 (4.86)
  Week 32 | 2.9 (4.27) | 1.4 (4.38)
  Week 36 | 2.6 (4.75) | 2.2 (3.55)
  Week 40 | 2.8 (5.98) | 2.2 (3.55)
  Week 44 | 1.8 (6.03) | 2.8 (5.10)
  Week 48 | 1.5 (3.66) | 1.4 (3.92)
  Week 52: number analyzed (Participants) | 7 | 12
  Week 52: number analyzed (eyes) | 7 | 16
  Week 52 | 0.9 (4.18) | 2.2 (3.30)
  Week 56 (Follow up): number analyzed (Participants) | 3 | 3
  Week 56 (Follow up): number analyzed (eyes) | 3 | 3
  Week 56 (Follow up) | 3.7 (5.67) | 1.6 (3.53)

31. Secondary Outcome: Open Label Extension Period: Visual Field Mean Deviation (dB) Measured by Humphrey From Baseline
Description: as for outcome 30
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160
Population: All participants for whom Visual Field Mean Deviation (dB) measured by Humphrey from Baseline was measured.
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
dB
  Week 68 | 3.3 (5.59) | 4.0 (6.66)
  Week 84 | 5.1 (6.66) | 4.4 (6.53)
  Week 100: number analyzed (Participants) | 8 | 11
  Week 100: number analyzed (eyes) | 8 | 14
  Week 100 | 3.1 (6.85) | 5.5 (8.04)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | 0.9 (0.97) | 2.9 (0.99)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | 4.4 (5.48) | 4.7 (6.21)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | 4.7 (8.43) | 4.0 (6.62)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | 5.5 (8.16) | 5.6 (9.51)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | 6.3 (13.67) | 11.5 (16.98)

32. Secondary Outcome: Double Masked Period: Color Discrimination - Number of Plates
Description: Double Masked Period: Change from Baseline in Color Discrimination - Number of Plates from Baseline by Visit by Ishihara Test. Score range: 0-38. Higher number equals better color discrimination equals better outcome. Lower number equals worse color discrimination equals worse outcome.
Time Frame: Assessed at each visit from Baseline to Week 56 (follow-up visit)
Population: All participants for whom Number of Plates was measured
Measure: Mean (Standard Deviation); unit: Plates
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
Plates
  Day 5 | 0.0 (0.00) | 0.1 (0.57)
  Week 4 | 0.0 (0.00) | 0.1 (0.50)
  Week 8 | 0.1 (0.35) | 0.3 (0.58)
  Week 12 | 0.3 (0.71) | 0.2 (0.75)
  Week 16 | 0.0 (0.00) | 0.4 (0.89)
  Week 20 | 0.5 (0.93) | 0.3 (0.60)
  Week 24 | 0.3 (0.71) | 0.5 (0.97)
  Week 28 | 0.9 (1.36) | 0.8 (1.39)
  Week 32 | 0.8 (1.16) | 0.7 (1.30)
  Week 36 | 0.8 (1.16) | 0.8 (1.05)
  Week 40 | 0.5 (0.76) | 0.6 (0.81)
  Week 44 | 1.0 (1.07) | 0.9 (1.31)
  Week 48 | 1.3 (1.39) | 1.1 (1.34)
  Week 52 | 1.6 (1.60) | 1.1 (1.09)
  Week 56 (Follow up): number analyzed (Participants) | 3 | 3
  Week 56 (Follow up): number analyzed (eyes) | 3 | 3
  Week 56 (Follow up) | 1.7 (2.89) | 1.0 (1.00)

33. Secondary Outcome: Open Label Extension Period: Change From Baseline in Color Discrimination - Number of Plates by Visit
Description: Open Label Extension Period: Change from Baseline in Color Discrimination - Number of Plates from Baseline by Visit by Ishihara Test. Score range: 0-38. Higher number equals better color discrimination equals better outcome. Lower number equals worse color discrimination equals worse outcome.
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160
Population: All participants for whom Color Discrimination - Number of Plates by Visit was measured.
Measure: Mean (Standard Deviation); unit: plates
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
plates
  Week 68 | 1.3 (1.28) | 1.4 (1.36)
  Week 84 | 1.9 (1.96) | 1.6 (1.75)
  Week 100: number analyzed (Participants) | 8 | 11
  Week 100: number analyzed (eyes) | 8 | 14
  Week 100 | 2.8 (3.65) | 2.0 (2.54)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | 0.0 (0.00) | 0.5 (0.71)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | 2.4 (2.70) | 1.2 (1.92)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | 2.0 (1.83) | 1.6 (1.33)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | 1.0 (0.82) | 0.9 (0.35)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | 2.0 (2.00) | 1.3 (1.53)

34. Secondary Outcome: Double Masked Period: Change From Baseline in Contrast Sensitivity by Pelli-Robson Contrast Sensitivity Chart by Visit
Description: Letters are arranged on a 60 x 85 cm chart in sets of triplets which contain the same contrast, decreasing in log10 contrast from top to bottom and left to right as participant progresses from one triplet to the other. Each group of three letters is decreased in contrast by a factor 0.71 (1/√2) (log contrast 0.15) of the proceeding set. Participant reads letters, starting with highest contrast, until unable to read letters in a single group. Score is based on the contrast of the last group read correctly.The size of the letters on the chart subtend 0.5 degrees at 3m, The test is scored in LogCS units, where each set of triplets advances in steps of 0.15 log units ranging from LogCS of 0.00 (approx. 100% contrast) to LogCS 2.25 (approx. 0.56% contrast). Change from baseline: the more negative the number means poor outcome, the more positive the number means better outcome.
Time Frame: Assessed at each visit from Baseline to Week 56 (follow-up visit)
Population: All participants for whom Contrast sensitivity was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
score on a scale
  Day 5 | 0.075 (0.0802) | -0.019 (0.1078)
  Week 4 | 0.038 (0.0694) | -0.028 (0.1366)
  Week 8 | 0.075 (0.1134) | 0.047 (0.1420)
  Week 12 | 0.056 (0.1116) | 0.000 (0.1342)
  Week 16 | 0.075 (0.1134) | -0.009 (0.1020)
  Week 20 | 0.094 (0.1116) | -0.009 (0.1020)
  Week 24 | 0.075 (0.1134) | 0.028 (0.1663)
  Week 28 | 0.113 (0.1747) | -0.009 (0.1393)
  Week 32 | 0.113 (0.1553) | 0.028 (0.1663)
  Week 36 | 0.150 (0.1604) | 0.056 (0.1806)
  Week 40 | 0.206 (0.1782) | 0.075 (0.1975)
  Week 44 | 0.225 (0.2268) | 0.066 (0.2625)
  Week 48 | 0.188 (0.2232) | 0.084 (0.1446)
  Week 52 | 0.225 (0.2121) | 0.075 (0.2258)
  Week 56 (Follow up): number analyzed (Participants) | 3 | 3
  Week 56 (Follow up): number analyzed (eyes) | 3 | 3
  Week 56 (Follow up) | 0.100 (0.0866) | 0.050 (0.0866)

35. Secondary Outcome: Open Label Extension Period: Change From Baseline in Contrast Sensitivity by Visit
Description: Letters are arranged on a 60 x 85 cm chart in sets of triplets which contain the same contrast, decreasing in log10 contrast from top to bottom and left to right as participant progresses from one triplet to the other. Each group of three letters is decreased in contrast by a factor 0.71 (1/√2) (log contrast 0.15) of the proceeding set. Participant reads letters, starting with highest contrast, until unable to read letters in a single group. Score is based on the contrast of the last group read correctly. The size of the letters on the chart subtend 0.5 degrees at 3m, The test is scored in LogCS units, where each set of triplets advances in steps of 0.15 log units ranging from LogCS of 0.00 (approx. 100% contrast) to LogCS 2.25 (approx. 0.56% contrast). Change from baseline: the more negative the number means poor outcome, the more positive the number means better outcome.
Time Frame: Assessed at each visit from Baseline from Week 68 to Week 160
Population: All participants for whom Contrast Sensitivity was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
score on a scale
  Week 68 | 0.225 (0.2121) | 0.084 (0.1972)
  Week 84 | 0.300 (0.1964) | 0.122 (0.1991)
  Week 100: number analyzed (Participants) | 8 | 11
  Week 100: number analyzed (eyes) | 8 | 14
  Week 100 | 0.281 (0.2034) | 0.118 (0.2893)
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104: number analyzed (eyes) | 2 | 2
  Week 104 | 0.075 (0.1061) | 0.075 (0.1061)
  Week 116: number analyzed (Participants) | 7 | 10
  Week 116: number analyzed (eyes) | 7 | 13
  Week 116 | 0.300 (0.3000) | 0.196 (0.2626)
  Week 132: number analyzed (Participants) | 7 | 10
  Week 132: number analyzed (eyes) | 7 | 13
  Week 132 | 0.214 (0.1909) | 0.127 (0.2796)
  Week 148: number analyzed (Participants) | 4 | 6
  Week 148: number analyzed (eyes) | 4 | 8
  Week 148 | 0.225 (0.2598) | 0.113 (0.1553)
  Week 160: number analyzed (Participants) | 3 | 3
  Week 160: number analyzed (eyes) | 3 | 3
  Week 160 | 0.150 (0.2598) | 0.100 (0.0866)

36. Secondary Outcome: Double Masked Change From Baseline in Retinal Ganglion Cell Layer Thickness
Description: Change from baseline in Retinal Ganglion Cell Layer Thickness by SD-OCT From Baseline by Visit
Time Frame: Assessed at Baseline and Week 52 (end-of-treatment visit)
Population: All participants for whom Retinal Ganglion Cell Layer Thickness was measured.
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
µm | -1.5 (4.00) | -3.6 (13.49)

37. Secondary Outcome: Open Label Extension Period: Change From Baseline in Retinal Ganglion Cell Layer Thickness
Description: Open Label Extension Period: Change from baseline in Retinal Ganglion Cell Layer Thickness by SD-OCT by SD-OCT by visit
Time Frame: Assessed at Baseline, Week 148,
Population: All participants for whom Change from baseline in Retinal Ganglion Cell Layer Thickness by SD-OCT was measured.
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 1 | 3
Number analyzed (eyes) | 1 | 5
µm | -1.0 | 3.4 (6.07)

38. Secondary Outcome: Double Masked: VFQ-39 Distance Activities Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Distance Activities score. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom VFQ-39 Distance Activities was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 9.4 (12.94) | 0.0 (14.03)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | 54.2 (14.43) |

39. Secondary Outcome: Open Label Extension Period: VFQ-39 Distance Activities Score
Description: Change in Visual Function Questionnaire (VFQ-39) Distance Activities Score.National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change in Visual Function Questionnaire (VFQ-39) Distance Activities score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 3
score on a scale | 12.5 (20.56) | 13.9 (6.36)

40. Secondary Outcome: Open Label Extension Period: VFQ-39 Social Functioning Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Social Functioning Score. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change in Visual Function Questionnaire (VFQ-39) Social Functioning score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 6
score on a scale | 8.3 (11.78) | 5.6 (17.35)

41. Secondary Outcome: Double Masked: VFQ-39 Social Functioning Score.
Description: as for outcome 40
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom VFQ-39 Social Functioning was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 6.3 (10.68) | 0.0 (19.25)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | 16.7 (8.34) |

42. Secondary Outcome: Double Masked: VFQ-39 Mental Health Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Mental Health score. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom VFQ-39 Mental Health was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 12.0 (9.16) | 19.7 (32.47)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | 13.3 (25.17) |

43. Secondary Outcome: Open Label Extension Period: VFQ-39 Mental Health Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Mental Health Score . National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change in Visual Function Questionnaire (VFQ-39) Mental Health score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 3
score on a scale | 16.4 (22.31) | 29.2 (29.83)

44. Secondary Outcome: Double Masked: VFQ-39 Role Difficulties Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Role Difficulties score National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom VFQ-39 Role Difficulties was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 4.7 (10.43) | 14.1 (9.38)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | 10.4 (13.01) |

45. Secondary Outcome: Open Label Extension Period: VFQ-39 Role Difficulties Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Role Difficulties Score. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change in Visual Function Questionnaire (VFQ-39) Role Difficulties score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 6
score on a scale | 8.0 (12.87) | 37.5 (16.54)

46. Secondary Outcome: Open Label Extension Period:VFQ-39 Dependency Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39 ) Dependency Score. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change in Visual Function Questionnaire (VFQ-39) Dependency Score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 6
score on a scale | 16.1 (13.91) | 27.1 (3.61)

47. Secondary Outcome: Double Masked: VFQ-39 Dependency Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Dependency score. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom VFQ-39 Dependency score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 9.4 (22.10) | -2.6 (24.85)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | -8.3 (23.66) |

48. Secondary Outcome: Double Masked: VFQ-39 Color Vision Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Color Vision score. National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom VFQ-39 Color Vision score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 6.3 (17.68) | 6.3 (12.50)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | 0.0 (25.00) |

49. Secondary Outcome: Open Label Extension Period: VFQ-39 Color Vision Score
Description: as for outcome 48
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change in Visual Function Questionnaire (VFQ-39) Color Vision Score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 6
score on a scale | -7.1 (18.90) | 8.3 (14.43)

50. Secondary Outcome: Double Masked: VFQ-39 Peripheral Score
Description: Change from baseline in Visual Function Questionnaire (VFQ-39) Peripheral Score . National Eye Institute VFQ-39 score measures health-related quality of life of subjects with visual impairment, in 12 domains: general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision and 1 composite score. Each domain is converted to a 0 to 100 scale; the lowest and highest possible scores are set at 0 and 100 points, respectively. Higher score means higher functioning. Scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. For the composite score, the vision-targeted sub-scale scores are averaged, excluding the general health questions. Domain scores from each cohort are averaged and the change from baseline per domain is calculated.
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom VFQ-39 Peripheral score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | 0.0 (13.36) | 6.3 (12.50)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | 66.7 (14.43) |

51. Secondary Outcome: Open Label Extension Period: Visual Function Questionnaire (VFQ-39) Peripheral Score
Description: as for outcome 50
Time Frame: Assessed at Baseline, Week 160 (End of OLE Period)
Population: All participants for whom Change in Visual Function Questionnaire (VFQ-39) Peripheral Score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye in DM Period | Bilateral Eye in DM Period
Number analyzed (Participants) | 7 | 3
Number analyzed (eyes) | 7 | 3
score on a scale | 0.0 (32.27) | 0.0 (25.00)

52. Secondary Outcome: Double Masked Period: Change in Intraocular Pressure (IOP)
Description: Double Masked Period: Change in intraocular Pressure (IOP) in mmHg from Baseline by Visit
Time Frame: as for outcome 1
Population: All participants for whom intraocular Pressure (IOP) was measured
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Double Masked Group Vehicle Eyes | Double Masked Group Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
mmHg
  Day 5 | -0.3 (1.67) | -0.2 (1.87)
  Week 4 | 0.0 (3.16) | -0.4 (2.16)
  Week 8 | -0.4 (1.77) | -0.5 (1.83)
  Week 12 | 0.5 (2.39) | -0.5 (2.53)
  Week 16 | 0.4 (1.51) | 0.6 (3.14)
  Week 20 | 0.4 (1.85) | -0.3 (1.66)
  Week 24 | -0.1 (3.31) | -0.4 (2.99)
  Week 28 | 0.3 (1.83) | 0.3 (1.88)
  Week 32 | 0.0 (2.62) | -0.3 (1.92)
  Week 36 | -1.1 (1.55) | -1.3 (1.96)
  Week 40 | 0.3 (2.25) | -0.6 (1.75)
  Week 44 | -0.4 (2.00) | -0.3 (1.85)
  Week 48 | 0.5 (3.66) | 0.8 (2.79)
  Week 52 | -1.0 (1.20) | -0.5 (2.66)
  Week 56 (follow up Visit) | -1.0 (1.20) | -0.5 (2.66)

53. Secondary Outcome: Open Label Extension Period: Intraocular Pressure (IOP)
Description: Change from baseline in Intraocular Pressure (IOP) in mmHg by Visit.
Time Frame: Assessed at Baseline, Week 68, 84, 100, 116, 132, 148, 152, Week 160/ (End of treatment visit)
Population: All participants for whom intraocular pressure was measured.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Vehicle to Elamipretide Eyes | Elamipretide to Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
Number analyzed (eyes) | 8 | 16
mmHg
  Week 68 | -0.4 (1.60) | 0.8 (2.49)
  Week 84 | 1.4 (3.29) | 0.4 (2.37)
  Week 100 | -0.9 (2.03) | -0.2 (2.22)
  Week 104 | 1.5 (2.12) | -1.0 (1.41)
  Week 116 | 0.1 (3.18) | -0.5 (2.63)
  Week 132 | 0.1 (1.35) | 0.1 (1.80)
  Week 148 | 1.3 (2.06) | -0.1 (2.36)
  Week 160 | 0.7 (0.58) | -1.7 (1.53)

54. Secondary Outcome: OLE: Slit Lamp Examination (SLE)-Vehicle Eye
Description: Open Label Extension: Shift in Slit Lamp Examination from Baseline by Visit: number of eyes that changed from normal or abnormal not clinically significant, to abnormal clinically significant for Vehicle Eyes
Time Frame: Assessed at Baseline, Week 68, 84, 100, 116, 132, 148, 152, Week 160/ (End of treatment visit)
Population: All participants for who SLE was measured.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Groups:
- Normal to Abnormal CS: Number of eyes shifting from normal to Abnormal clinically significant in slit lamp findings
- Shift From Abnormal NCS to Abnormal CS: Number of eyes shifting from Abnormal nonclinically significant to abnormal clinically significant
Arm/Group | Normal to Abnormal CS | Shift From Abnormal NCS to Abnormal CS
Number analyzed (Participants) | 8 | 8
Number analyzed (Eyes) | 8 | 8
eyes
  Lids Eye Week 68 | 0 | 0
  Lids Week 84 | 0 | 0
  Lids Week 100 | 0 | 0
  Lids Week 104: number analyzed (Participants) | 2 | 2
  Lids Week 104: number analyzed (Eyes) | 2 | 2
  Lids Week 104 | 0 | 0
  Lids Week 116: number analyzed (Participants) | 7 | 7
  Lids Week 116: number analyzed (Eyes) | 7 | 7
  Lids Week 116 | 0 | 0
  Lids Week 132: number analyzed (Participants) | 7 | 7
  Lids Week 132: number analyzed (Eyes) | 7 | 7
  Lids Week 132 | 0 | 0
  Lids Week 148: number analyzed (Participants) | 4 | 4
  Lids Week 148: number analyzed (Eyes) | 4 | 4
  Lids Week 148 | 0 | 0
  Lids Week 160: number analyzed (Participants) | 3 | 3
  Lids Week 160: number analyzed (Eyes) | 3 | 3
  Lids Week 160 | 0 | 0
  Conjunctiva 68 | 0 | 0
  Conjunctiva 84 | 0 | 0
  Conjunctiva 100 | 0 | 0
  Conjunctiva 104: number analyzed (Participants) | 2 | 2
  Conjunctiva 104: number analyzed (Eyes) | 2 | 2
  Conjunctiva 104 | 0 | 0
  Conjunctiva 116: number analyzed (Participants) | 7 | 7
  Conjunctiva 116: number analyzed (Eyes) | 7 | 7
  Conjunctiva 116 | 0 | 0
  Conjunctiva 132: number analyzed (Participants) | 7 | 7
  Conjunctiva 132: number analyzed (Eyes) | 7 | 7
  Conjunctiva 132 | 0 | 0
  Conjunctiva 148: number analyzed (Participants) | 4 | 4
  Conjunctiva 148: number analyzed (Eyes) | 4 | 4
  Conjunctiva 148 | 0 | 0
  Conjunctiva 160: number analyzed (Participants) | 3 | 3
  Conjunctiva 160: number analyzed (Eyes) | 3 | 3
  Conjunctiva 160 | 0 | 0
  Cornea Week 68 | 0 | 0
  Cornea Week 84 | 1 | 0
  Cornea Week 100 | 1 | 0
  Cornea Week 104: number analyzed (Participants) | 2 | 2
  Cornea Week 104: number analyzed (Eyes) | 2 | 2
  Cornea Week 104 | 0 | 0
  Cornea Week 116: number analyzed (Participants) | 7 | 7
  Cornea Week 116: number analyzed (Eyes) | 7 | 7
  Cornea Week 116 | 0 | 0
  Cornea Week 132: number analyzed (Participants) | 7 | 7
  Cornea Week 132: number analyzed (Eyes) | 7 | 7
  Cornea Week 132 | 0 | 0
  Cornea Week 148: number analyzed (Participants) | 4 | 4
  Cornea Week 148: number analyzed (Eyes) | 4 | 4
  Cornea Week 148 | 0 | 0
  Cornea Week 160: number analyzed (Participants) | 3 | 3
  Cornea Week 160: number analyzed (Eyes) | 3 | 3
  Cornea Week 160 | 0 | 0
  Anterior Chamber 68 | 0 | 0
  Anterior Chamber 84 | 0 | 0
  Anterior Chamber 100 | 0 | 0
  Anterior Chamber 104: number analyzed (Participants) | 2 | 2
  Anterior Chamber 104: number analyzed (Eyes) | 2 | 2
  Anterior Chamber 104 | 0 | 0
  Anterior Chamber 116: number analyzed (Participants) | 7 | 7
  Anterior Chamber 116: number analyzed (Eyes) | 7 | 7
  Anterior Chamber 116 | 0 | 0
  Anterior Chamber 132 | 0 | 0
  Anterior Chamber 148: number analyzed (Participants) | 4 | 4
  Anterior Chamber 148: number analyzed (Eyes) | 4 | 4
  Anterior Chamber 148 | 0 | 0
  Anterior Chamber 160: number analyzed (Participants) | 3 | 3
  Anterior Chamber 160: number analyzed (Eyes) | 3 | 3
  Anterior Chamber 160 | 0 | 0
  Iris Week 68 | 0 | 0
  Iris Week 84 | 0 | 0
  Iris Week 100 | 0 | 0
  Iris Week 104: number analyzed (Participants) | 2 | 2
  Iris Week 104: number analyzed (Eyes) | 2 | 2
  Iris Week 104 | 0 | 0
  Iris Week 116: number analyzed (Participants) | 7 | 7
  Iris Week 116: number analyzed (Eyes) | 7 | 7
  Iris Week 116 | 0 | 0
  Iris Week 132: number analyzed (Participants) | 7 | 7
  Iris Week 132: number analyzed (Eyes) | 7 | 7
  Iris Week 132 | 0 | 0
  Iris Week 148: number analyzed (Participants) | 8 | 7
  Iris Week 148: number analyzed (Eyes) | 8 | 7
  Iris Week 148 | 0 | 0
  Iris Week 160 | 0 | 0
  Lens Week 68 | 0 | 0
  Lens Week 84 | 0 | 0
  Lens Week 100 | 0 | 0
  Lens Week 104: number analyzed (Participants) | 2 | 2
  Lens Week 104: number analyzed (Eyes) | 2 | 2
  Lens Week 104 | 0 | 0
  Lens Week 116: number analyzed (Participants) | 7 | 7
  Lens Week 116: number analyzed (Eyes) | 7 | 7
  Lens Week 116 | 1 | 0
  Lens Week 132: number analyzed (Participants) | 7 | 7
  Lens Week 132: number analyzed (Eyes) | 7 | 7
  Lens Week 132 | 0 | 0
  Lens Week 148: number analyzed (Participants) | 4 | 4
  Lens Week 148: number analyzed (Eyes) | 4 | 4
  Lens Week 148 | 0 | 0
  Lens Week 160: number analyzed (Participants) | 3 | 3
  Lens Week 160: number analyzed (Eyes) | 3 | 3
  Lens Week 160 | 0 | 0
  Vitreous Week 68 | 0 | 0
  Vitreous Week 84 | 0 | 0
  Vitreous Week 100 | 0 | 0
  Vitreous Week 104: number analyzed (Participants) | 2 | 2
  Vitreous Week 104: number analyzed (Eyes) | 2 | 2
  Vitreous Week 104 | 0 | 0
  Vitreous Week 116: number analyzed (Participants) | 7 | 7
  Vitreous Week 116: number analyzed (Eyes) | 7 | 7
  Vitreous Week 116 | 0 | 0
  Vitreous Week 132: number analyzed (Participants) | 7 | 7
  Vitreous Week 132: number analyzed (Eyes) | 7 | 7
  Vitreous Week 132 | 0 | 0
  Vitreous Week 148: number analyzed (Participants) | 4 | 4
  Vitreous Week 148: number analyzed (Eyes) | 4 | 4
  Vitreous Week 148 | 0 | 0
  Vitreous Week 160: number analyzed (Participants) | 3 | 3
  Vitreous Week 160: number analyzed (Eyes) | 3 | 3
  Vitreous Week 160 | 0 | 0
  Retina Week 68 | 0 | 0
  Retina Week 84 | 0 | 0
  Retina Week 100 | 0 | 0
  Retina Week 104: number analyzed (Participants) | 2 | 2
  Retina Week 104: number analyzed (Eyes) | 2 | 2
  Retina Week 104 | 0 | 0
  Retina Week 116: number analyzed (Participants) | 7 | 7
  Retina Week 116: number analyzed (Eyes) | 7 | 7
  Retina Week 116 | 0 | 0
  Retina Week 132: number analyzed (Participants) | 7 | 7
  Retina Week 132: number analyzed (Eyes) | 7 | 7
  Retina Week 132 | 0 | 0
  Retina Week 148: number analyzed (Participants) | 4 | 4
  Retina Week 148: number analyzed (Eyes) | 4 | 4
  Retina Week 148 | 0 | 0
  Retina Week 160: number analyzed (Participants) | 3 | 3
  Retina Week 160: number analyzed (Eyes) | 3 | 3
  Retina Week 160 | 0 | 0
  Optic nerve Week 68 | 0 | 0
  Optic nerve Week 84 | 0 | 0
  Optic nerve Week 100 | 0 | 0
  Optic nerve Week 104: number analyzed (Participants) | 2 | 2
  Optic nerve Week 104: number analyzed (Eyes) | 2 | 2
  Optic nerve Week 104 | 0 | 0
  Optic nerve Week 116: number analyzed (Participants) | 7 | 7
  Optic nerve Week 116: number analyzed (Eyes) | 7 | 7
  Optic nerve Week 116 | 0 | 0
  Optic nerve Week132: number analyzed (Participants) | 7 | 7
  Optic nerve Week132: number analyzed (Eyes) | 7 | 7
  Optic nerve Week132 | 0 | 0
  Optic nerve Week 148: number analyzed (Participants) | 4 | 4
  Optic nerve Week 148: number analyzed (Eyes) | 4 | 4
  Optic nerve Week 148 | 0 | 0
  Optic nerve Week 160: number analyzed (Participants) | 3 | 3
  Optic nerve Week 160: number analyzed (Eyes) | 3 | 3
  Optic nerve Week 160 | 0 | 0
  Macula Week 68 | 0 | 0
  Macula Week 84 | 0 | 0
  Macula Week 100 | 0 | 0
  Macula Week 104: number analyzed (Participants) | 2 | 2
  Macula Week 104: number analyzed (Eyes) | 2 | 2
  Macula Week 104 | 0 | 0
  Macula Week 116: number analyzed (Participants) | 7 | 7
  Macula Week 116: number analyzed (Eyes) | 7 | 7
  Macula Week 116 | 0 | 0
  Macula Week 132: number analyzed (Participants) | 7 | 7
  Macula Week 132: number analyzed (Eyes) | 7 | 7
  Macula Week 132 | 0 | 0
  Macula Week 148: number analyzed (Participants) | 4 | 4
  Macula Week 148: number analyzed (Eyes) | 4 | 4
  Macula Week 148 | 0 | 0
  Macula Week 160: number analyzed (Participants) | 3 | 3
  Macula Week 160: number analyzed (Eyes) | 3 | 3
  Macula Week 160 | 0 | 0
  Choroid Week 68 | 0 | 0
  Choroid Week 84 | 0 | 0
  Choroid Week 100 | 0 | 0
  Choroid Week 104: number analyzed (Participants) | 2 | 2
  Choroid Week 104: number analyzed (Eyes) | 2 | 2
  Choroid Week 104 | 0 | 0
  Choroid Week 116: number analyzed (Participants) | 7 | 7
  Choroid Week 116: number analyzed (Eyes) | 7 | 7
  Choroid Week 116 | 0 | 0
  Choroid Week 132: number analyzed (Participants) | 7 | 7
  Choroid Week 132: number analyzed (Eyes) | 7 | 7
  Choroid Week 132 | 0 | 0
  Choroid Week 148: number analyzed (Participants) | 4 | 4
  Choroid Week 148: number analyzed (Eyes) | 4 | 4
  Choroid Week 148 | 0 | 0
  Choroid Week 160: number analyzed (Participants) | 3 | 3
  Choroid Week 160: number analyzed (Eyes) | 3 | 3
  Choroid Week 160 | 0 | 0
  Periphery Week 68 | 0 | 0
  Periphery Week 84 | 0 | 0
  Periphery Week 100 | 0 | 0
  Periphery Week 104: number analyzed (Participants) | 2 | 2
  Periphery Week 104: number analyzed (Eyes) | 2 | 2
  Periphery Week 104 | 0 | 0
  Periphery Week 116: number analyzed (Participants) | 7 | 7
  Periphery Week 116: number analyzed (Eyes) | 7 | 7
  Periphery Week 116 | 0 | 0
  Periphery Week 132: number analyzed (Participants) | 7 | 7
  Periphery Week 132: number analyzed (Eyes) | 7 | 7
  Periphery Week 132 | 0 | 0
  Periphery Week 148: number analyzed (Participants) | 4 | 4
  Periphery Week 148: number analyzed (Eyes) | 4 | 4
  Periphery Week 148 | 0 | 0
  Periphery 160: number analyzed (Participants) | 3 | 3
  Periphery 160: number analyzed (Eyes) | 3 | 3
  Periphery 160 | 0 | 0

55. Secondary Outcome: OLE: Slit Lamp Examination (SLE)-Elamipretide Eye
Description: Open Label Extension: Shift in Slit Lamp Examination from Baseline by Visit: number of eyes that changed from normal or abnormal not clinically significant, to abnormal clinically significant for Elamipretide Eyes
Time Frame: Assessed at Baseline, Week 68, 84, 100, 116, 132, 148, 152, Week 160/ (End of treatment visit)
Population: All participants for who SLE was measured.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Normal to Abnormal CS | Shift From Abnormal NCS to Abnormal CS
Number analyzed (Participants) | 12 | 12
Number analyzed (Eyes) | 16 | 16
eyes
  Lids Eye Week 68 | 0 | 0
  Lids Week 84 | 0 | 0
  Lids Week 100: number analyzed (Eyes) | 14 | 14
  Lids Week 100 | 0 | 0
  Lids Week 104: number analyzed (Eyes) | 2 | 2
  Lids Week 104 | 0 | 0
  Lids Week 116: number analyzed (Eyes) | 13 | 13
  Lids Week 116 | 0 | 0
  Lids Week 132: number analyzed (Eyes) | 13 | 13
  Lids Week 132 | 0 | 0
  Lids Week 148: number analyzed (Eyes) | 8 | 8
  Lids Week 148 | 0 | 0
  Lids Week 160: number analyzed (Eyes) | 3 | 3
  Lids Week 160 | 0 | 0
  Conjunctiva 68 | 0 | 0
  Conjunctiva 84 | 0 | 0
  Conjunctiva 100: number analyzed (Eyes) | 14 | 14
  Conjunctiva 100 | 0 | 0
  Conjunctiva 104: number analyzed (Eyes) | 2 | 2
  Conjunctiva 104 | 0 | 0
  Conjunctiva 116: number analyzed (Eyes) | 13 | 13
  Conjunctiva 116 | 0 | 0
  Conjunctiva 132: number analyzed (Eyes) | 13 | 13
  Conjunctiva 132 | 0 | 0
  Conjunctiva 148: number analyzed (Eyes) | 8 | 8
  Conjunctiva 148 | 0 | 0
  Conjunctiva 160: number analyzed (Eyes) | 3 | 3
  Conjunctiva 160 | 0 | 0
  Cornea Week 68 | 0 | 0
  Cornea Week 84 | 0 | 0
  Cornea Week 100: number analyzed (Eyes) | 14 | 14
  Cornea Week 100 | 0 | 0
  Cornea Week 104: number analyzed (Eyes) | 2 | 2
  Cornea Week 104 | 0 | 0
  Cornea Week 116: number analyzed (Eyes) | 13 | 13
  Cornea Week 116 | 0 | 0
  Cornea Week 132: number analyzed (Eyes) | 13 | 13
  Cornea Week 132 | 0 | 0
  Cornea Week 148: number analyzed (Eyes) | 8 | 8
  Cornea Week 148 | 0 | 0
  Cornea Week 160: number analyzed (Eyes) | 3 | 3
  Cornea Week 160 | 0 | 0
  Anterior Chamber 68 | 0 | 0
  Anterior Chamber 84 | 0 | 0
  Anterior Chamber 100: number analyzed (Eyes) | 14 | 14
  Anterior Chamber 100 | 0 | 0
  Anterior Chamber 104: number analyzed (Eyes) | 2 | 2
  Anterior Chamber 104 | 0 | 0
  Anterior Chamber 116: number analyzed (Eyes) | 13 | 13
  Anterior Chamber 116 | 0 | 0
  Anterior Chamber 132: number analyzed (Eyes) | 13 | 13
  Anterior Chamber 132 | 0 | 0
  Anterior Chamber 148: number analyzed (Eyes) | 8 | 8
  Anterior Chamber 148 | 0 | 0
  Anterior Chamber 160: number analyzed (Eyes) | 3 | 3
  Anterior Chamber 160 | 0 | 0
  Iris Week 68 | 0 | 0
  Iris Week 84 | 0 | 0
  Iris Week 100: number analyzed (Eyes) | 14 | 14
  Iris Week 100 | 0 | 0
  Iris Week 104: number analyzed (Eyes) | 2 | 2
  Iris Week 104 | 0 | 0
  Iris Week 116: number analyzed (Eyes) | 13 | 13
  Iris Week 116 | 0 | 0
  Iris Week 132: number analyzed (Eyes) | 13 | 13
  Iris Week 132 | 0 | 0
  Iris Week 148: number analyzed (Eyes) | 8 | 8
  Iris Week 148 | 0 | 0
  Iris Week 160: number analyzed (Eyes) | 3 | 3
  Iris Week 160 | 0 | 0
  Lens Week 68 | 0 | 0
  Lens Week 84 | 0 | 0
  Lens Week 100: number analyzed (Eyes) | 8 | 8
  Lens Week 100 | 0 | 0
  Lens Week 104: number analyzed (Eyes) | 2 | 2
  Lens Week 104 | 0 | 0
  Lens Week 116: number analyzed (Eyes) | 13 | 13
  Lens Week 116 | 1 | 0
  Lens Week 132: number analyzed (Eyes) | 13 | 13
  Lens Week 132 | 0 | 0
  Lens Week 148: number analyzed (Eyes) | 8 | 8
  Lens Week 148 | 0 | 0
  Lens Week 160: number analyzed (Eyes) | 3 | 3
  Lens Week 160 | 0 | 0
  Vitreous Week 68 | 0 | 0
  Vitreous Week 84 | 0 | 0
  Vitreous Week 100: number analyzed (Eyes) | 14 | 14
  Vitreous Week 100 | 0 | 0
  Vitreous Week 104: number analyzed (Eyes) | 2 | 2
  Vitreous Week 104 | 0 | 0
  Vitreous Week 116: number analyzed (Eyes) | 13 | 13
  Vitreous Week 116 | 0 | 0
  Vitreous Week 132: number analyzed (Eyes) | 13 | 13
  Vitreous Week 132 | 0 | 0
  Vitreous Week 148: number analyzed (Eyes) | 8 | 8
  Vitreous Week 148 | 0 | 0
  Vitreous Week 160: number analyzed (Eyes) | 3 | 3
  Vitreous Week 160 | 0 | 0
  Retina Week 68 | 0 | 0
  Retina Week 84 | 0 | 0
  Retina Week 100: number analyzed (Eyes) | 14 | 14
  Retina Week 100 | 0 | 0
  Retina Week 104: number analyzed (Eyes) | 2 | 2
  Retina Week 104 | 0 | 0
  Retina Week 116: number analyzed (Eyes) | 13 | 13
  Retina Week 116 | 0 | 0
  Retina Week 132: number analyzed (Eyes) | 13 | 13
  Retina Week 132 | 0 | 0
  Retina Week 148: number analyzed (Eyes) | 8 | 8
  Retina Week 148 | 0 | 0
  Retina Week 160: number analyzed (Eyes) | 3 | 3
  Retina Week 160 | 0 | 0
  Optic nerve Week 68 | 0 | 0
  Optic nerve Week 84 | 0 | 0
  Optic nerve Week 100: number analyzed (Eyes) | 14 | 14
  Optic nerve Week 100 | 0 | 0
  Optic nerve Week 104: number analyzed (Eyes) | 2 | 2
  Optic nerve Week 104 | 0 | 0
  Optic nerve Week 116: number analyzed (Eyes) | 13 | 13
  Optic nerve Week 116 | 0 | 0
  Optic nerve Week 132: number analyzed (Eyes) | 13 | 13
  Optic nerve Week 132 | 0 | 0
  Optic nerve Week 148: number analyzed (Eyes) | 8 | 8
  Optic nerve Week 148 | 0 | 0
  Optic nerve Week 160: number analyzed (Eyes) | 3 | 3
  Optic nerve Week 160 | 0 | 0
  Macula Week 68 | 0 | 0
  Macula Week 84 | 0 | 0
  Macula Week 100: number analyzed (Eyes) | 14 | 14
  Macula Week 100 | 0 | 0
  Macula Week 104: number analyzed (Eyes) | 2 | 2
  Macula Week 104 | 0 | 0
  Macula Week 116: number analyzed (Eyes) | 13 | 13
  Macula Week 116 | 0 | 0
  Macula Week 132: number analyzed (Eyes) | 13 | 13
  Macula Week 132 | 0 | 0
  Macula Week 148: number analyzed (Eyes) | 8 | 8
  Macula Week 148 | 0 | 0
  Macula Week 160: number analyzed (Eyes) | 3 | 3
  Macula Week 160 | 0 | 0
  Choroid Week 68 | 0 | 0
  Choroid Week 84 | 0 | 0
  Choroid Week 100: number analyzed (Eyes) | 14 | 14
  Choroid Week 100 | 0 | 0
  Choroid Week 104: number analyzed (Eyes) | 2 | 2
  Choroid Week 104 | 0 | 0
  Choroid Week 116: number analyzed (Eyes) | 13 | 13
  Choroid Week 116 | 0 | 0
  Choroid Week 132: number analyzed (Eyes) | 13 | 13
  Choroid Week 132 | 0 | 0
  Choroid Week 148: number analyzed (Eyes) | 8 | 8
  Choroid Week 148 | 0 | 0
  Choroid Week 160: number analyzed (Eyes) | 3 | 3
  Choroid Week 160 | 0 | 0
  Periphery Week 68 | 0 | 0
  Periphery Week 84 | 0 | 0
  Periphery Week 100: number analyzed (Eyes) | 14 | 14
  Periphery Week 100 | 0 | 0
  Periphery Week 104: number analyzed (Eyes) | 2 | 2
  Periphery Week 104 | 0 | 0
  Periphery Week 116: number analyzed (Eyes) | 13 | 13
  Periphery Week 116 | 0 | 0
  Periphery Week 132: number analyzed (Eyes) | 13 | 13
  Periphery Week 132 | 0 | 0
  Periphery Week 148: number analyzed (Eyes) | 8 | 8
  Periphery Week 148 | 0 | 0
  Periphery 160: number analyzed (Participants) | 3 | 12
  Periphery 160: number analyzed (Eyes) | 3 | 3
  Periphery 160 | 0 | 0

56. Secondary Outcome: Double Masked: Slit Lamp Changes From Baseline: Vehicle Eye and Elamipretide Eye
Description: Incidence of Change from normal or Abnormal, clinically insignificant to normal clinically significant
Time Frame: as for outcome 1
Measure: Number; unit: eyes
Arm/Group | Double Masked Group Vehicle Eyes | Double Masked Group Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
eyes
  Conjunctiva Week 4 Normal to Abnormal Clinically significant | 1 | 0
  Conjunctiva: Week 8 Normal to Abnormal Clinically significant | 1 | 0
  Conjunctiva: Week 16 Normal to Abnormal Clinically significant | 1 | 1
  Conjunctiva: Week 28 Normal to Abnormal Clinically significant | 1 | 1
  Conjunctiva: Week 44 Normal to Abnormal Clinically significant | 1 | 1
  Lids: Week 28 Normal to Abnormal Clinically significant | 0 | 1
  Cornea: Week 32 Normal to Abnormal Clinically significant | 0 | 2
  Cornea: Week 44 Normal to Abnormal Clinically significant | 1 | 1

57. Secondary Outcome: Double Masked: Dilated Fundus Changes From Baseline: Vehicle Eye and Elamipretide Eyes
Description: Double Masked: Dilated Fundus Changes from Baseline: Vehicle Eye and Elamipretide Eyes Incidence of Change from normal or Abnormal-clinically insignificant, to normal clinically significant
Time Frame: as for outcome 1
Population: All participants for whom dilated fundus was measured.
Measure: Number; unit: eyes
Groups:
- Vehicle Eyes: Vehicle Eyes: Number of eyes shifting from normal or Abnormal- non clinically significant, to Abnormal clinically significant
- Elamipretide Eyes: Elamipretide Eyes: Number of eyes shifting from normal or Abnormal-non clinically significant, to abnormal clinically significant
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 12
eyes | 0 | 0

58. Secondary Outcome: Open Label Extension Period: Dilated Fundus Changes From Baseline: Vehicle Eye and Elamipretide Eyes
Description: Incidence of Change from normal or Abnormal-clinically insignificant, to normal clinically significant
Time Frame: Assessed at Baseline, Week 68, 84, 100, 116, 132, 148, 152, Week 160/ (End of treatment visit)
Population: All participants for whom dilated fundus was measured.
Measure: Number; unit: eyes
Arm/Group | Vehicle Eyes | Elamipretide Eyes
Number analyzed (Participants) | 8 | 16
eyes | 0 | 0

59. Secondary Outcome: Double Masked: VFQ-39 General Health Score
Description: as for outcome 21
Time Frame: Assessed at Baseline, Week 52 (end-of-treatment visit) and Week 56 (follow-up visit)
Population: All participants for whom VFQ-39 General Health score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Single Eye | Bilateral Eye
Number analyzed (Participants) | 8 | 4
Number analyzed (eyes) | 8 | 8
score on a scale
  Week 52 | -3.8 (10.09) | -0.6 (19.72)
  Week 56 (Follow-up Visit): number analyzed (Participants) | 3 | 0
  Week 56 (Follow-up Visit): number analyzed (eyes) | 3 | 0
  Week 56 (Follow-up Visit) | -5.8 (6.29) |

ADVERSE EVENTS:
Time Frame: Up to 112 weeks
Groups:
- One Eye DM Period: One eye Double Masked (DM) Period One drop elamipretide (MTP-131) 1% topical ophthalmic solution BID applied to a single eye and one drop of vehicle topical ophthalmic solution BID in the fellow eye
- Both Eyes DM Period: Both eyes Double Masked (DM) One drop elamipretide (MTP-131) 1% topical ophthalmic solution BID applied to both eyes (OU).
- (One Eye DM Period) OLE: Both eyes Open label Extension period One drop elamipretide (MTP-131) 1% topical ophthalmic solution BID applied to both eyes (OU) (and one eye in DM period)
- (Both Eyes DM) OLE Period: Both eyes Open label Extension period One drop elamipretide (MTP-131) 1% topical ophthalmic solution BID applied to both eyes (OU) (and both eyes in DM period)
Arm/Group | One Eye DM Period | Both Eyes DM Period | (One Eye DM Period) OLE | (Both Eyes DM) OLE Period
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 6/8 | 3/4 | 7/8 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | One Eye DM Period (N=8) | Both Eyes DM Period (N=4) | (One Eye DM Period) OLE (N=8) | (Both Eyes DM) OLE Period (N=4)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 2 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 3 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT02693119/Prot_SAP_000.pdf